CLINICAL TRIAL: NCT05236725
Title: Systematic Monitoring and Remote Testing of Blood Pressure in Postpartum Women
Brief Title: Monitoring and Testing of Blood Pressure in Postpartum Women
Acronym: SMART-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00077904
Record Dates: First submitted 2022-01-28; First posted 2022-02-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: postpartum; blood pressure; women; blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Subjects randomized to SOC arm are provided with the appropriate standard of care depending upon their risk level (as determined by their individual provider or WFBMC Maternal-Fetal Medicine provider)
- Remote Blood Pressure Monitoring (rBPM) (Experimental): Subjects randomized to rBPM arm receive the appropriate standard of care depending upon their risk level, as well as the remote BP monitoring app (BabyScripts) and Bluetooth enabled BP cuff/monitor, and will receive the following equipment and monitoring:
  * a specialized, Bluetooth enabled BP monitoring cuff (Clinically Validated, A&D Medical Wireless Blood Pressure Monitor-Upper Arm (Appendix 2)
  * BP monitoring smart phone app, BabyScripts™
  * Verbal and written instructions, to conduct BP checks at home
  Interventions: Device: Remote Blood Pressure Cuff; Device: Blood Pressure (BP) monitoring smart phone app, BabyScripts™; Behavioral: Instructions

INTERVENTIONS:
Device: Remote Blood Pressure Cuff — specialized, Bluetooth enabled BP monitoring cuff
  Arms: Remote Blood Pressure Monitoring (rBPM)
Device: Blood Pressure (BP) monitoring smart phone app, BabyScripts™ — app that works with the monitoring cuff
  Arms: Remote Blood Pressure Monitoring (rBPM)
Behavioral: Instructions — Verbal and written instructions to conduct BP checks at home
  Arms: Remote Blood Pressure Monitoring (rBPM)

SUMMARY:
The purpose of this research study is to find out the usefulness of checking a woman's blood pressure remotely (at home) for 3 weeks after being discharged from the hospital after having a baby (or babies). Some women can develop hypertension, or high BP, after delivery even if they have not had this problem before or during their pregnancy. Untreated or unknown high BP can lead to medical complications, and if severe, can be life threatening. Monitoring, or checking, remote BP after a woman has delivered her baby (or babies) has been suggested to be a better way to monitor BPs without having to stay in the hospital for a longer time after delivery. Other researchers report that women who have checked their BP remotely after delivery found out that this was both possible and acceptable.

DETAILED DESCRIPTION:
This is a randomized control trial (RCT). All women, 18 years of age and older, delivering an infant(s) at The Birth Center at Atrium Health Wake Forest Baptist and residing in Forsyth County, NC that have been approached by our Home Visit Coordinators will be eligible for enrollment and invited to participate in the SMART- BP study prior to discharge from the postpartum unit. Per established protocols, the Home Visit Coordinators for the Nurse Education Support Team Program attempt to approach all women that deliver in The Birth Center and who reside in Forsyth County. At this initial introduction, the Home Visit Coordinators determine if the patient has any need for, or interest in, any of the vetted community resources available to her and her family. Information about any of these resources are provided to the patient at that time. Additionally, the Home Visit Coordinators offer to schedule a nurse "home visit". This nurse home visit occurs via phone call, telehealth visit, or an in person visit ~2 weeks after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women that received prenatal care at one of the Atrium Health Wake Forest Baptist OB/MFM outpatient clinic locations in Forsyth County, NC
* Women that delivered an infant(s) at The Birth Center at Atrium Health Wake Forest Baptist
* Women that delivered an infant(s) at home or outside facility, and were transported to Atrium Health Wake Forest Baptist and received postpartum care in The Birth Center
* Currently resides in Forsyth County, NC
* 18 years of age or older
* Able to read and understand either English or Spanish
* Owns or has daily access to a smart phone (iOS or Android operating system) with available Wi-Fi or monthly mobile data plan

Exclusion Criteria:

* Women that received postpartum care at any location other than The Birth Center at Atrium Health Wake Forest Baptist
* Resides outside of Forsyth County, NC
* Under 18 years of age
* Unable to read or understand either English or Spanish
* Does not own or have daily access to a smart phone (iOS or Android operating system) with available Wi-Fi or monthly mobile data plan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1602 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Median number of rBPM measures obtained | Discharge through Week 3 postpartum
  Used to determine feasibility of remote blood pressure monitoring intervention (rBPM)
Proportion of women monitoring blood pressure (BP) according to American College of Obstetricians and Gynecologists (ACOG) guidelines | Day 10 postpartum
  Impact of rBPM on adherence to ACOG recommendations
Median total cost of health care | From discharge through week 8 postpartum
Median number of Severe Hypertension events | Discharge through week 1 postpartum
Median number of Severe Hypertension events | Discharge through week 3 postpartum
Median number of encounters for urgent or emergent care | Discharge through week 3 postpartum
  Study team will use the electronic health record to identify encounters to the Emergency Department, OB Triage, and Urgent Care facilities

SECONDARY OUTCOMES:
Median number of encounters for urgent or emergent care | Discharge through week 8 postpartum
  Study team will use the electronic health record to identify encounters to the Emergency Department, OB Triage, and Urgent Care facilities
Acceptability of rBPM in postpartum period | Week 3 postpartum
  Survey to determine subject's level of satisfaction with use of the rBPM tools. Survey responses will be compared among subjects from varying demographic and socioeconomic groups. Survey is designed utilizing a Likert-type scale with 1-2 being higher level of acceptability, 3 being neutral, and 4-5 being lower level of acceptability of the rBPM tools. Study team will report the overall proportion and estimate the proportion of women with higher vs. lower levels of acceptability among women of different demographic and socioeconomic groups. This aim only applies to the women in the treatment (rBPM) arm.
Median Length of Stay (LOS) in hospital after delivery | Baseline (date of delivery) through discharge, assessed for up to 8 weeks postpartum
Median number of hospital readmissions | Discharge through week 8 postpartum
Median Length of Stay (LOS) for hospital readmissions | Discharge through week 8 postpartum
Median number of women that have a follow-up encounter scheduled with their Primary Care Physician (PCP) within 12 months after delivery | Discharge through 12 months postpartum

OTHER OUTCOMES:
Validate and calibrate previously developed predictive algorithm | Discharge through week 8 postpartum
  Intended to assess the performance of the predictive algorithm in identifying postpartum high blood pressure readmissions. Study team will utilize blood pressure measures obtained through 3 weeks postpartum, as well as any hypertensive disorders of pregnancy events postpartum through 8 weeks postpartum, to include ED/Urgent Care/OB Triage encounters and any readmissions. The predictive algorithm is informed by information documented in the electronic health record, prior to delivery and during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth T Jensen, MPH PhD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05236725/ICF_000.pdf